CLINICAL TRIAL: NCT00750802
Title: A Phase 1, Single Centre, Single Dose, Double-Blind, Double-Dummy, Four-Way Crossover, Placebo-Controlled, Randomized Study to Investigate the Effects of AZD6280 on Sedation, Cognition and EEG in Comparison With Lorazepam in Healthy Male Volunteers
Brief Title: A Sedation/Cognition/EEG Study Using AZD6280 and Comparator
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Mark Smith, MD, MSD, Emerging Psychiatry, AstraZeneca Pharmaceuticals
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: D0850C00014; Eudract # 2008-001757-17
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2009-06-26 (Estimated); Status verified 2009-06

CONDITIONS: Healthy Volunteer
Keywords: Phase I
MeSH Terms: interventions — 4-amino-8-(2,5-dimethoxyphenyl)-N-propylcinnoline-3-carboxamide; Lorazepam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Experimental)
  Interventions: Drug: AZD6280
- 2 (Experimental)
  Interventions: Drug: AZD6280
- 3 (Active Comparator)
  Interventions: Drug: Lorazepam
- 4 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD6280 — 10mg Capsule, oral, single-dose
  Arms: 1
Drug: AZD6280 — 40mg Capsule, oral, single-dose
  Arms: 2
Drug: Lorazepam — 2mg tablet, oral single-dose
  Other Names: Ativan
  Arms: 3
Drug: Placebo
  Arms: 4

SUMMARY:
The purpose of the study is to determine the effects of AZD6280 compared to lorazepam on sleepiness, concentration and brain activity.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and female subjects aged 18 to 55 years (inclusive) on Day 1.
* Female subjects must be of non-child bearing potential.

Exclusion Criteria:

* Clinically significant illness within 2 weeks before the study start.
* Enrollment in another concurrent investigational study or intake of an investigational drug within 30 days or intake of an investigational drug within a period of 5 half lives of that drug prior to the screening visit
* Blood loss in excess of 200 mL within 30 days of Day -2, in excess of 400 mL within 90 days of Day -2, or in excess of 1200 mL within 1 year of Day -2
* Clinically relevant abnormalities in physical examinations, vital signs, ECG, clinical chemistry, hematology or urinalysis

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2008-09; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Evaluation of the pharmacodynamic effects of AZD6280 by central nervous system function tests | Test batteries will be performed at specified times both before and following study drug administration

SECONDARY OUTCOMES:
Evaluation and characterization of the pharmacokinetics of AZD6280 | Blood samples will be taken during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Leiden, Netherlands